CLINICAL TRIAL: NCT05529771
Title: Clinical Outcomes of paTients pREsenting to HArare COVID-19 CenTer of Excellence With SARS-CoV-2 Infection - (TREAT Study)
Brief Title: Clinical Outcomes of paTients pREsenting to HArare COVID-19 CenTer of Excellence With SARS-CoV-2 Infection
Acronym: TREAT
Status: Completed | Type: Observational
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: UNITAID (Other)
Responsible Party: Sponsor
Other Study IDs: EG0281
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: COVID-19
Keywords: Antigen rapid diagnostic test; COVID-19; Health Facilities; Africa
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In order to influence COVID-19 treatment guidelines, evidence on disease progression and clinical outcomes of hospitalized COVID-19 patients, particularly those receiving innovative COVID-19 medications in an African setting is critical. This study will be conducted by EGPAF to describe patient characteristics, COVID-19 illness progression, and clinical outcomes among hospitalized COVID-19 patients at Parirenyatwa General and Harare Teaching Hospitals, COVID Centers of Excellence at in Zimbabwe.

DETAILED DESCRIPTION:
Rationale:

Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a novel coronavirus first identified in December of 2019 in Wuhan, China. Since the first case of COVID-19 was diagnosed in 2019, the number of cases has exponentially increased globally. As of December 16th 2021, there have been over 270 million confirmed cases of COVID-19 and over 5.3 million deaths from COVID-19 across the world. Zimbabwe is one of the countries in Southern Africa affected by the COVID-19 pandemic. World Health Organization (WHO) recommended treatment with IL-6 receptor blockers for patients with severe or critical COVID-19 disease in addition to the previous recommendation of systemic corticosteroids.

Primary objectives

1. To describe the clinical course and outcomes of patients admitted to the Harare Teaching Hospital - Parirenyatwa General Hospital with SARS-CoV-2 infection.

   1. Clinical course includes disease severity, use of oxygen, ICU admission, mechanical ventilation, treatments received, and duration of care.
   2. Outcomes include death, discharged or still hospitalized.
   3. Among discharged, outcomes will include readmission, persistent symptoms or recovery at 3 months post diagnosis.
2. To determine individual-level factors associated with clinical course and disease outcome including but not limited to demographics, population (healthy adults, children, pregnant women), comorbidities (i.e. HIV, TB, diabetes, cardiovascular disease [CVD], obesity), SARS-CoV-2 vaccine status, lab/medical history, COVID-19 treatment, and disease severity at presentation.

Secondary objective

1. To document pharmacovigilance around the use of new COVID-19 treatments, including side effects and any associated treatment interruptions.

Design: We propose an observational cohort study with a retrospective and a prospective component to collect data on patients admitted to Parirenyatwa and Harare Hospitals with SARS-CoV-2 infection for COVID-19 care. Retrospective review and abstraction of information from medical records will be conducted on all COVID-19 admissions from January 2022 to July/August 2022 depending on when all approvals are in place to initiate primary data collection. Subsequently, the study team will enroll participants through March 2023 and prospectively follow all admitted COVID-19 patients until they meet a clinical outcome (death, discharge) up to 3 months after SARS-CoV-2 diagnosis. Data on disease progression, need for oxygen, ICU care or mechanical ventilation, treatments received, treatment side effects, laboratory results, duration of hospitalization and outcome (death, discharge or still hospitalized) will be abstracted from all patient medical records. For patients enrolled in the prospective cohort, a detailed medical and SARS-CoV-2 related history will be collected at the admission to the hospital. In addition, study staff will conduct short telephone interviews with study participants to document their course at home after discharge.

ELIGIBILITY:
Inclusion criteria:

* Patient admitted with documented SARS-CoV-2 infection.
* Willing and able to provide written informed consent or parental consent (with assent if applicable) for the prospective study cohort.

Exclusion criteria:

• None.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to the study facility for COVID-19 care and treatment during the study period regardless of age or disease state. A sample size of approximately 400 participants is estimated to be included, but could be fewer or higher number of participants depending on the stage of the pandemic.
Sampling Method: Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Disease severity | 3 months
  Number of patients died, discharged, or still hospitalized, as a proportion of patients admitted with COVID-19 disease
Discharged patients | 3 months
  Number of patients readmitted, experiencing persistent symptoms, recovered, as a proportion of patients admitted with COVID-19 disease

SECONDARY OUTCOMES:
COVID-19 Treatment Pharmacovigilance | 3 months
  Types of side effects, and/or any associated treatment interruptions

CONTACTS AND LOCATIONS:
Overall Officials: Nilesh Bhatt, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation; Simba Mashizha, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (1):
- Parirenyatwa General Hospital, Harare, Zimbabwe